CLINICAL TRIAL: NCT01898026
Title: Development of Palatable Soluble Fibre Containing Carbohydrate Foods and Its Effects on Postprandial Blood Glucose Response in Healthy Individuals
Brief Title: Soluble Fibre Enriched CHO Food Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Principal Investigator, Vladimir Vuksan, Professor, Unity Health Toronto
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: White Line; 12-379C (Other: St. Michael's Hospital Research Ethics Board)
Record Dates: First submitted 2013-07-09; First posted 2013-07-12 (Estimated); Last update posted 2014-02-05 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes; Healthy
Keywords: PGX; fibre; postprandial glycemia
MeSH Terms: conditions — Diabetes Mellitus | interventions — Bread

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PGX (Experimental): samples of white bread, mashed potatoes, muffin, hot breakfast cereal with the addition of soluble fibre blend
  Interventions: Dietary Supplement: Bread; Dietary Supplement: Mashed Potatoes; Dietary Supplement: Muffins; Dietary Supplement: Hot Breakfast Cereal
- Control (Other): samples of white bread, mashed potatoes, muffin, hot breakfast cereal without the addition of soluble fibre blend
  Interventions: Dietary Supplement: Bread; Dietary Supplement: Mashed Potatoes; Dietary Supplement: Muffins; Dietary Supplement: Hot Breakfast Cereal

INTERVENTIONS:
Dietary Supplement: Bread — Samples of white bread, with or without the addition of PGX fibre blend
Dietary Supplement: Mashed Potatoes — samples of mashed potatoes, with or without the addition of soluble fibre blend
Dietary Supplement: Muffins — Samples of muffins, with or without the addition of PGX fibre blend
Dietary Supplement: Hot Breakfast Cereal — Samples of hot breakfast cereal without the addition of soluble fibre blend

SUMMARY:
The proposed study will examine the effects of incorporating a soluble fibre blend into commonly consumed refined carbohydrate foods on sensory parameters and postprandial blood glucose. A sensory evaluation will be conducted in phase I to asses for differences between the control and fibre enriched samples of white bread, mashed potatoes, muffin, hot breakfast cereal. Phase II will be investigating the postprandial blood glucose responses of the 8 test foods from phase I.

DETAILED DESCRIPTION:
Literature to date points to beneficial glycemic effects from consumption of soluble fibre; however, whole grain products consumption is below recommendations possibly due to the presence of unappealing characteristic organoleptic properties. White, refined products are still the choice of the general public. As such, we propose to investigate the feasibility of increasing health benefits of commonly consumed white, refined carbohydrate products by incorporating a soluble fibre blend.

This research is important to determine the feasibility of developing fibre enriched carbohydrate foods that maintains the original organoleptic properties and is effective in reducing postprandial blood glucose response.

35 subjects will be recruited in phase I to complete a sensory evaluation on the test foods. Following tasting of the control and fibre-enriched samples, data on each subjects' liking or disliking will be collected through a 9-point hedonic scale.

An acute crossover RCT will be conducted in phase II by 10 healthy individuals. Subjects will be randomized to consume one the treatments at each visit and blood glucose levels over 120min and satiety scores will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Normotensive (SBP<140mmHg, DBP <90mmHg)
* BMI 18.5 - 25 kg/m2
* Post-menopausal or not pregnant women

Exclusion Criteria:

* Allergy or sensitivity to test meals
* Swallowing difficulties
* Chronic use of medications or fibre
* GI conditions affecting stomach pH
* Must not be enrolled in another study
* History of liver or kidney disease, diabetes, hypertension, stroke or myocardial infarctions, thyroid disease, celiac /gastrointestinal disease, HIV positive or AIDS

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Sensory Evaluation | 1 month
  Subjects will be recruited in phase I to complete a sensory evaluation on the test foods. Following tasting of the control and fibre-enriched samples, data on each subjects' liking or disliking will be collected through a 9-point hedonic scale.
Postprandial Glycemia | 3 months
  Subjects will be randomized to consume one of the 8 interventions at each visit and blood glucose levels over 120min and satiety scores will be measured.

SECONDARY OUTCOMES:
Satiety Score | 3 months
  The incorporation of viscous soluble fibre in commonly consumed carbohydrate foods will result in increase in subjective satiety compared to non soluble fibre enriched products. Satiety will be measured using a satiety questionnaire in which you will answer four questions about how full you feel.

OTHER OUTCOMES:
Safety | 3 montsh
  Safety will monitored using a symptoms questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — St. Michael's & University of Toronto
Locations (1):
- St. Michael's, Toronto, Ontario, Canada